CLINICAL TRIAL: NCT07135466
Title: A Phase 1/2 Study of T-cell Expressing an Anti-CD22 Chimeric-Antigen Receptor (SHB-04-CD22) in Patients With CD22-expressing B-cell Malignancies
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Elad Jacoby, MD, Principal Investigator, Pediatric Hematology and Oncology, Sheba Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHB-04-CD22; 2289-25-SMC (Other: EC identifier)
Record Dates: First submitted 2025-07-02; First posted 2025-08-22 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: B Cell Malignancies
Keywords: ALL; NHL; DLBCL; CAR-T; CD22; Chimeric Antigen Receptor; Leukemia; Lymphoma
MeSH Terms: conditions — Leukemia; Lymphoma

STUDY DESIGN:
Intervention Model Description: Single arm, open label, non-randomized trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm, open label, dose escalation: Anti CD22 CAR-T (SHB-04-CD22) (Experimental): Phase 1 of this study includes a dose escalation plan of anti CD22 CAR-T (SHB-04-CD22). Treatment will start at dose level 1. According to safety assessments, dose will increase to next dose level.
  Dose level 1: 3x10^5 CAR+ T cells per kilogram Dose level 2: 1x10^6 CAR+ T cells per kilogram Dose level 3: 3x10^6 CAR+ T cells per kilogram
  Phase 2 of this study will be a dose expansion phase of the dose recommended based on safety and expected efficacy.
  Interventions: Other: CD22 CAR-T cells

INTERVENTIONS:
Other: CD22 CAR-T cells — CD22 CAR-T cells

SUMMARY:
This is a phase I/II trial of T-cell expressing an anti-CD22 Chimeric-Antigen-Receptor (CAR) in patients with CD22 expressing B-cell malignancies. This trial is an open label, single-arm, for pediatric and adult patients with relapsed/refractory B-cell malignancies.

DETAILED DESCRIPTION:
B-cell precursor Acute Lymphoblastic Leukemia (ALL) is the most common pediatric cancer, and an adult malignancy with poor prognosis. B-cell non-Hodgkin lymphoma (NHL) and common lymphocytic leukemia (CLL) arise from mature B-cells, and are more commonly seen in the adult and elderly population. In the recent decade, advances in immunotherapy targeting cell surface markers, using antibodies, antibody-drug conjugates, bispecific antibodies or CAR-T cells, have improved the outcome of patients with relapsed and refractory B-cell malignancies. CAR-T cell products targeting CD19, a common B-cell antigen, are approved for B-cell malignancies. Treatment with CD19 CAR-T cells was FDA approved for pediatric ALL, adult ALL, diffuse large B-cell lymphoma (DLBCL), follicular lymphoma, mantle-cell lymphoma (MCL) and primary mediastinal B-cell lymphoma (PMBCL). Still, most patients with B-cell malignancies treated nowadays with commercial CD19 CAR T-cells relapse. To address this, alternative immunotherapy targets have been proposed. CD22 is an additional co-receptor on B-cells, commonly expressed in B-cell malignancies such as ALL, and has been most studied in this context. Autologous T cells will be harvested from patients with B-cell malignancies and then activated and transduced with a retrovirus containing a chimeric-antigen receptor (CAR), manufactured by the Advanced Biotherapy Center (ABC) at the Sheba Medical Center. Patients will undergo a one-time cell collection via apheresis, after which the cells will be sent to the laboratory for activation and introduction of a gene that recognizes the CD22 antigen. Patients will receive lymphodepleting chemotherapy followed by a single dose of CD22 CAR-T cells (SHB-04-CD22), after which they will be monitored and undergo various research assessments (including blood tests, genetic tests, and assessments of the disease status). Patients will be closely monitored for approximately 3 months after treatment to assess response and safety of the treatment. Long-term survival monitoring will take place once a year for 15 years.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have a CD22-expressing hematologic malignancy, relapsed or refractory after receiving at least 2 lines of standard therapy including CD19-directed therapy (For CD19 positive disease):
* Relapse following standard relapse protocol (2nd relapse), including CD19 CART.
* Primary refractory, i.e. failed to achieve morphologic remission after 2 lines of induction chemotherapy.
* Age 1-80 years
* CD22 expression shown by flow cytometry on at least 70% of leukemic blasts / lymphoma cells
* Adequate CD3 count (above 120 CD3+ cells per microliter blood)
* Clinical performance status: Patients > 10 years of age: Karnofsky ≥ 50%; Patients ≤ 10 years of age: Lansky scale ≥ 50%. Exception for neurologic symptoms (e.g. paralysis) that are explained by the malignancy.
* Females of child-bearing potential must have a negative pregnancy test
* Cardiac function: LV ejection fraction >45% or shortening fraction >28%
* At least 60 days after autologous or allogeneic BMT
* At least 30 days after prior CAR therapy in absence of response

Ages: 1 Year to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-04-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Safety Evaluation: Treatment Related Toxicities | From enrollment to 3 months post treatment.
  An evaluation of safety of the use of autologous anti-CD22 CAR T cells (SHB-04-CD22) manufactured at the Sheba Medical Center, in patients with relapsed/refractory B-cell malignancies. Safety will be determined by evaluation of participants with treatment-related adverse events, as assessed by CTCAE 5.0.
Efficacy Evaluation | 1 month to 1 year post treatment.
  An evaluation of the feasibility and efficacy of administering anti-CD22-CAR T cells (SHB-04-CD22) in patients with B-cell malignancies at the Sheba Medical Center. Efficacy will be determined by an evaluation of disease response in participants post treatment. Disease response will be assessed by blasts percentage in bone marrow for ALL patients and by PET-CT scan based on the Lugano classification for NHL patients.
Minimal toxic dose evaluation | From first dose to end 3 months post treatment.
  An evaluation of the minimal toxic dose of CD22 CAR-T cells (SHB-04-CD22). This will be determined by evaluation of participants with treatment-related adverse events, as assessed by CTCAE 5.0, and according to different dose levels administered.

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Elad Jacoby, MD, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba Medical Center, Ramat Gan, G, Israel

IPD SHARING:
Plan to Share IPD: Yes
Only IPD used in the results publication